CLINICAL TRIAL: NCT01746082
Title: A Phase II Open-Label Study in Healthy Adult and Elderly Populations to Assess the Safety, Reactogenicity, and Immunogenicity of an Intramuscular Unadjuvanted Subvirion Monovalent Inactivated Influenza H3N2 Variant (H3N2v) Vaccine
Brief Title: Safety and Immunogenicity of a Monovalent Inactivated Influenza H3N2 Variant (H3N2v) Vaccine in Adult and Elderly Populations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-0011; HHSN272200800002C
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-01

CONDITIONS: Influenza
Keywords: influenza, H3N2, H3N2v, vaccine, unadjuvanted, Parent Protocol
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- Subjects 18 - 64 years (Experimental): 100 (up to 120) subjects 18 - 64 years old receive two doses of monovalent inactivated influenza H3N2 variant (MIV), delivered intramuscularly as 15 micrograms (mcg) of hemagglutinin (HA)/0.5 milliliter (mL) dose, 21 days apart.
  Interventions: Biological: Influenza A/H3N2 variant Vaccine
- Subjects > /= 65 years (Experimental): 100 (up to 120) subjects greater than or equal to 65 years old receive two doses of monovalent inactivated influenza H3N2 variant (MIV), delivered intramuscularly as 15 micrograms (mcg) of hemagglutinin (HA)/0.5 milliliter (mL) dose, 21 days apart.
  Interventions: Biological: Influenza A/H3N2 variant Vaccine

INTERVENTIONS:
Biological: Influenza A/H3N2 variant Vaccine — Investigational influenza virus H3N2v vaccine, a monovalent type A inactivated vaccine (H3N2v MIV) for intramuscular use, is a sterile clear and slightly opalescent suspension prepared from influenza virus propagated in embryonated chicken eggs. The H3N2v MIV contains no preservative. Subjects will be stratified by age (approximately 100 (up to 120) subjects 18-64 years old and approximately 100 (up to 120) subjects >/=65 years old) to receive two doses of H3N2v MIV, delivered intramuscularly as 15 micrograms (mcg) of hemagglutinin (HA)/0.5 milliliter (mL) dose, 21 days apart

SUMMARY:
This is a Phase II open-label study in approximately 200, and up to 240, healthy males and non-pregnant females, aged 18 years and older. This study is designed to assess the safety, reactogenicity, and immunogenicity of an unadjuvanted subvirion monovalent inactivated influenza H3N2v vaccine manufactured by Sanofi Pasteur. Subjects will be stratified by age (approximately 100 (up to 120) subjects 18-64 years old and approximately 100 (up to 120) subjects >/= 65 years old) to receive two doses of vaccine, delivered intramuscularly as 15mcg HA/0.5mL dose, 21 days apart. The duration of the study for each subject will be approximately 7 months.

DETAILED DESCRIPTION:
This is a Phase II open-label study in approximately 200 (up to 240) healthy males and non-pregnant females, aged 18 years and older. This study is designed to assess the safety, reactogenicity, and immunogenicity of an unadjuvanted subvirion monovalent inactivated influenza H3N2 variant (H3N2v) vaccine (MIV) manufactured by Sanofi Pasteur. Subjects will be stratified by age (approximately 100 (up to 120) subjects 18-64 years old and approximately 100 (up to 120) subjects >/= 65 years old) to receive two doses of H3N2v MIV, delivered intramuscularly as 15 micrograms (mcg) of hemagglutinin (HA)/0.5 milliliter (mL) dose, 21 days apart (see Table 1). Subjects may receive licensed seasonal influenza vaccine prior to (2 weeks if given the inactivated vaccine or 4 weeks if given the live, attenuated vaccine) the first H3N2v vaccination. Alternatively, subjects may receive licensed seasonal influenza vaccine at any time after completion of the Day 42 visit or following an early termination visit. Safety will be measured by the occurrence of solicited injection site and systemic reactogenicity on the day of each H3N2v vaccination through 7 days after each H3N2v vaccination, adverse events through 42 days after the first H3N2v vaccination, and serious adverse events (SAEs) and new-onset chronic medical conditions through 7 months after the first H3N2v vaccination. Immunogenicity testing will include performing hemagglutination inhibition (HAI) and neutralizing (Neut) antibody assays on serum obtained on the day of and prior to each H3N2v vaccination (Days 0 and 21), approximately 8 days after each H3N2v vaccination (Days 8 and 29), and approximately 21 days after the second H3N2v vaccination (Day 42).

From a subset of healthy adult subjects (up to 30 volunteers 18-64 years old enrolled at the Emory VTEU site who consent to blood donation for the immunology exploratory assays), an additional volume of venous blood will be drawn on Days 0, 8, 21, 29 and 42 to determine the specificity/cross reactivity of antibodies from H3N2v-reactive B cells with other influenza subtypes (e.g., 2009 H1N1 pandemic HA) and most recent H3 seasonal HA to define the molecular profile of antibody repertoire changes in circulating B cells after H3N2v vaccination, and to characterize the antibody-secreting cell (ASC), monoclonal antibody (mAb), and CD4+ T cell responses to H3N2v vaccination. The duration of the study for each subject will be approximately 7 months. Parent protocol to sub-study 12-0089 and 12-0015.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Are males or non-pregnant females, aged 18 years or older, inclusive.
4. Are in good health, as determined by vital signs (oral temperature, pulse and blood pressure), medical history and targeted physical examination based on medical history to ensure any existing medical diagnoses or conditions are stable (Stable chronic medical condition - no change in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome will not be considered a violation of this inclusion criterion.) Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity. Note: Topical, nasal, and inhaled medications; vitamins; and contraceptives are permitted with the exception of high dose inhaled steroids (see exclusion criteria #13).
5. Oral temperature is less than 100.4°F.
6. Pulse is 50 to 100 bpm.
7. Systolic blood pressure is 90 to 150 mm Hg.
8. Diastolic blood pressure is 60 to 100 mmHg.
9. Women of childbearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who are not postmenopausal for greater than or equal to 1 year) must agree to practice adequate contraception (abstinence from sexual intercourse with men, monogamous relationship with a vasectomized partner who was vasectomized at least 6 months prior to the subject receiving the first H3N2v vaccination, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices NuvaRing®, successful Essure® placement (permanent, non-surgical, non-hormonal sterilization) with documented confirmation test at least 3 months after the procedure), licensed hormonal methods such as implants, injectables or oral contraceptives (the pill), and any other Food and Drug Administration (FDA) approved birth control method) for at least 30 days prior to the first H3N2v vaccination through at least 30 days after the last H3N2v vaccination . Method of contraception will be captured on the appropriate data collection form.
10. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to each H3N2v vaccination.

Exclusion Criteria:

1. Have an acute illness, including an oral temperature greater than or equal to 100.4°F, within 3 days prior to each H3N2v vaccination.
2. Have any condition that, in the opinion of the site principal investigator or appropriate sub-investigator, would place the subject at an unacceptable risk of injury, render them unable to meet the requirements of the protocol or confound the interpretation of results.
3. Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months.
4. Have known active neoplastic disease or a history of any hematologic malignancy.
5. Have known HIV, hepatitis B, or hepatitis C infection.
6. Have a known allergy to eggs, egg or chicken protein, or other components of the H3N2v MIV (including octylphenol ethoxylate (Triton® X-100), gelatin, formaldehyde, and phosphate buffered saline).
7. Have a history of severe reactions following previous immunization with licensed influenza virus vaccines.
8. Have a history of Guillain-Barre Syndrome.
9. Have a history of alcohol or drug abuse in the last 5 years.
10. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other major psychiatric diagnosis.
11. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others, within the past 10 years.
12. Have taken high dose oral or parenteral glucocorticoids for 2 weeks or more in total at any time during the past 2 months. High dose defined as prednisone greater than or equal to 20mg total daily dose, or equivalent dose of other glucocorticoids.
13. Have taken high-dose inhaled steroids within the past 4 weeks. High dose defined as >800mcg/day of beclomethasone dipropionate or equivalent.
14. Have taken systemic corticosteroids of any dose within the past 4 weeks.
15. Received any licensed live vaccine within 4 weeks or any licensed inactivated vaccine within 2 weeks prior to the first H3N2v vaccination or planned receipt of any vaccine within 42 days after the first H3N2v vaccination. This is inclusive of licensed seasonal influenza vaccines.
16. Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within the 3 months prior to each H3N2v vaccination.
17. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to the first H3N2v vaccination.
18. Are participating or plan to participate in another clinical trial with an interventional agent (licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication) during the 7-month study period.
19. Are enrolled or plan to enroll in another clinical trial that has a study intervention such as a drug, biologic, device, blood product, or medication that could interfere with the safety assessment of the investigational product at any time during the 7-month study period.
20. Participated in an influenza A/H3N2v vaccine study in the past in a group receiving vaccine (does not apply to documented placebo recipients) or have a history of A/H3N2v infection prior to enrollment.
21. Plan to travel outside the U.S. (continental U.S., Hawaii and Alaska) in the time between the first H3N2v vaccination and 42 days after the first H3N2v vaccination.
22. Women who are breastfeeding or plan to breastfeed at any given time during the 7-month study period.
23. Occupational exposure to or direct physical contact with pigs in the past year.
24. Blood donation within 30 days prior to enrollment (only for a subset of healthy adult subjects - up to 30 volunteers 18-64 years old enrolled at the Emory VTEU site who consent to blood donation for the immunology exploratory assays).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects, stratified by age, achieving seroconversion (defined as either a pre-vaccination HAI titer <1:10 and a post-vac. HAI titer >/= 1:40 or a pre-vac. HAI titer >/= 1:10 and a minimum four-fold rise in post-vac. HAI antibody titer). | 21 days following the first vaccination
Safety: Occurrence of solicited injection site and systemic reactogenicity on the day of each H3N2v vaccination through 7 days after each H3N2v vaccination. | Through Day 7 following each vaccination
Immunogenicity: Proportion of subjects, stratified by age, achieving a serum HAI antibody titer of 1:40 or greater approximately 21 days following receipt of the first dose of H3N2v MIV against the H3N2v antigen contained in the H3N2v MIV. | 21 days following the first vaccination
Safety: Occurrence of H3N2v MIV-related serious adverse events from the time of first H3N2v vaccination through 7 months after the first H3N2v vaccination. | Through 7 months following the first vaccination

SECONDARY OUTCOMES:
Percentage of subjects, stratified by age, achieving either a pre-vaccination Neut titer <1:10 and a post-vaccination Neut titer >/=1:40 or a pre-vaccination Neut titer >/=1:10 and a minimum four-fold rise in post-vaccination Neut antibody titer. | 8, 21, 29 and 42 days following the first vaccination
Immunogenicity: Proportion of subjects, stratified by age, achieving a serum HAI antibody titer of 1:40 or greater approximately 8, 29 and 42 days following receipt of the first dose of H3N2v MIV against the H3N2v antigen contained in the H3N2v MIV. | 8, 29 and 42 days following the first vaccination
Immunogenicity: Geometric Mean Titers of serum HAI and Neut antibody at baseline, and approximately 8, 21, 29 and 42 days after the first H3N2v vaccination. | Baseline, 8, 21, 29 and 42 days following the first vaccination
Percentage of subjects, stratified by age, achieving seroconversion (defined as either a pre-vaccination HAI titer <1:10 and a post-vac. HAI titer >/=1:40 or a pre-vac. HAI titer >/=1:10 and a minimum four-fold rise in post-vac. HAI antibody titer). | 8, 29 and 42 days following the first vaccination
Immunogenicity: Proportion of subjects, stratified by age, achieving a serum Neut antibody titer of 1:40 or greater approximately 8, 21, 29 and 42 days following receipt of the first dose of H3N2v MIV against the H3N2v antigen contained in the H3N2v MIV. | 8, 21, 29 and 42 days following the first vaccination

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - University of Iowa - Infectious Disease Clinic, Iowa City, Iowa
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - Group Health Research Institute - Seattle, Seattle, Washington

REFERENCES:
- [Derived] Keitel WA, Jackson LA, Edupuganti S, Winokur PL, Mulligan MJ, Thornburg NJ, Patel SM, Rouphael NG, Lai L, Bangaru S, McNeal MM, Bellamy AR, Hill HR; VTEU H3N2v Vaccine Study Work Group. Safety and Immunogenicity of a Subvirion Monovalent Unadjuvanted Inactivated Influenza A(H3N2) Variant Vaccine in Healthy Persons >/=18 Years Old. J Infect Dis. 2015 Aug 15;212(4):552-61. doi: 10.1093/infdis/jiv056. Epub 2015 Feb 3. PMID 25649171